CLINICAL TRIAL: NCT01745263
Title: Vitamin D3 - Omega3 - Home Exercise - Healthy Ageing and Longevity Trial (Acronym: DO-HEALTH)
Brief Title: DO-HEALTH / Vitamin D3 - Omega3 - Home Exercise - Healthy Ageing and Longevity Trial
Acronym: DO-HEALTH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Recruitment Partners (Unknown); University of Geneva, Switzerland (Other); University of Basel (Other); University Hospital, Toulouse, France (Prof. Bruno Vellas, MD) (Unknown); Charite University, Berlin, Germany (Other); Medical University Innsbruck (Other); University of Coimbra, Portugal (Prof. José daSilva, MD) (Unknown); Other University Partners (Unknown); University of Sheffield (Other); University of Manchester, UK (Prof. David Felson, MD MPH) (Unknown); Max Rubner University, Germany (Prof. Bernhard Watzl, PhD) (Unknown); Technische Universität Dresden (Other); Impact Partner (Unknown); International Osteoporosis Foundation (IOF; Prof. John Kanis, MD) (Unknown); SME Partners (Unknown); Ferrari Data Solution (Other); Gut Pictures, Switzerland (Benno Gut; animated exercise video) (Unknown); NOVAMEN, France (Sandrine Rival; logistic management partner) (Unknown); Pharmalys, UK (Marieme Ba; monitoring partner) (Unknown); Industry Partners (Unknown); DSM Nutritional Products (Dr. Elisabeth Stöcklin PhD, Dr. Manfred Eggersdorfer PhD) (Unknown); Nestlé (Michaela Höhne PhD, Irène Corthesy PhD) (Unknown); Roche Diagnostics GmbH (Industry); European Commission (Other); Further collaborators and advisors at website do-health.eu (Unknown)
Responsible Party: Principal Investigator, Heike Bischoff-Ferrari, Director, Centre on Aging and Mobility, University of Zurich
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KEK-ZH-2012-0249; DO-HEALTH (Other Grant/Funding Number: European Commission (project number 278588))
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Improve Healthy Ageing in Seniors; Prevent Disease at Older Age
MeSH Terms: interventions — Cholecalciferol; Fatty Acids, Omega-3; Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- VitD-Omega3-StrengthExercise (Active Comparator): Vitamin D3 (2000 IU/d); Omega-3 fatty acids (1 g/d); Strength Home Exercise (3*30 minutes/week)
  Interventions: Drug: Vitamin D3; Drug: Omega 3 fatty acids; Procedure: Strength Home Exercise
- VitD-Omega3-FlexibilityExercise (Active Comparator): Vitamin D3 (2000 IU/d); Omega-3 fatty acids (1 g/d); Flexibility Home Exercise (3*30 minutes/week)
  Interventions: Drug: Vitamin D3; Drug: Omega 3 fatty acids; Procedure: Flexibility Home Exercise
- Placebo-Omega3-StrengthExercise (Active Comparator): Placebo Vitamin D3; Omega-3 fatty acids (1 g/d); Strength Home Exercise (3*30 minutes/week)
  Interventions: Drug: Omega 3 fatty acids; Procedure: Strength Home Exercise
- Placebo-Omega3-FlexibilityExercise (Active Comparator): Placebo Vitamin D3; Omega-3 fatty acids (1 g/d); Flexibility Home Exercise (3*30 minutes/week)
  Interventions: Drug: Omega 3 fatty acids; Procedure: Flexibility Home Exercise
- VitD-Placebo-StrengthExercise (Active Comparator): Vitamin D3 (2000 IU/d); Placebo Omega-3 fatty acids; Strength Home Exercise (3*30 minutes/week)
  Interventions: Drug: Vitamin D3; Procedure: Strength Home Exercise
- VitD-Placebo-FlexiblityExercise (Active Comparator): Vitamin D3 (2000 IU/d); Placebo Omega-3 fatty acids; Flexibility Home Exercise (3*30 minutes/week)
  Interventions: Drug: Vitamin D3; Procedure: Flexibility Home Exercise
- Placebo-Placebo-StrengthExercise (Active Comparator): Placebo Vitamin D3; Placebo Omega-3 fatty acids; Strength Home Exercise (3*30 minutes/week)
  Interventions: Procedure: Strength Home Exercise
- Placebo-Placebo-FlexibilityExercise (Sham Comparator): Placebo Vitamin D3; Placebo Omega-3 fatty acids; Flexibility Home Exercise (3*30 minutes/week)
  Interventions: Procedure: Flexibility Home Exercise

INTERVENTIONS:
Drug: Vitamin D3 — 2000 IU/d
  Other Names: Cholecalciferol
  Arms: VitD-Omega3-FlexibilityExercise; VitD-Omega3-StrengthExercise; VitD-Placebo-FlexiblityExercise; VitD-Placebo-StrengthExercise
Drug: Omega 3 fatty acids — Ratio EPA:DHA = 1:2
  1 g/d
  Other Names: Eicosapentaenoic acid AND Docosahexaenoic acid
  Arms: Placebo-Omega3-FlexibilityExercise; Placebo-Omega3-StrengthExercise; VitD-Omega3-FlexibilityExercise; VitD-Omega3-StrengthExercise
Procedure: Strength Home Exercise
  Arms: Placebo-Omega3-StrengthExercise; Placebo-Placebo-StrengthExercise; VitD-Omega3-StrengthExercise; VitD-Placebo-StrengthExercise
Procedure: Flexibility Home Exercise
  Arms: Placebo-Omega3-FlexibilityExercise; Placebo-Placebo-FlexibilityExercise; VitD-Omega3-FlexibilityExercise; VitD-Placebo-FlexiblityExercise

SUMMARY:
The European population is aging rapidly which poses a challenge on the individual, the European societies, and health care systems. Among the most promising public health interventions that may extend healthy life expectancy at older age are vitamin D, marine omega-3 fatty acids and physical exercise. However, their individual and combined effects have yet to be confirmed in a clinical trial.

The broad aim of DO-HEALTH is to prolong healthy life expectancy in European seniors. The specific aim is to establish whether vitamin D, omega-3 fatty acids, and a simple home exercise program will prevent disease at older age.

To achieve these aims, DO-HEALTH will enroll 2152 community-dwelling men and women who are 70 years and older, an age when chronic diseases increase substantially. The DO-HEALTH seniors will be recruited from 7 European cities (Zurich, Basel, Geneva, Toulouse, Berlin, Innsbruck and Coimbra) and will be randomized in a 2x2x2 factorial design trial to a simple home exercise program and/or vitamin D, and/or omega-3 fatty acids, over a 3 year period. This will allow to test the individual and the combined benefit of the interventions in the prevention of 5 primary endpoints: incident non-vertebral fractures; functional decline; systolic and diastolic blood pressure change; cognitive decline; and the rate of any infection. Key secondary endpoints include incidence of hip fractures, rate of falls, severity of pain in symptomatic knee osteoarthritis, gastro-intestinal symptoms, mental and oral health, quality of life, and mortality.

All clinical endpoints will be supported by a large DO-HEALTH biomarker study to evaluate the effect of the interventions at the cellular level of multi-organ function. DO-HEALTH will further evaluate reasons why or why not seniors adhere to the 3 interventions, and will assess their cost-benefit in a health economic model based on documented health care utilization and observed incidence of chronic disease.

website DO-HEALTH: http://do-health.eu/wordpress/

DETAILED DESCRIPTION:
The 3 primary treatment comparisons are:

1. 2000 IU vitamin D per day compared to placebo (controlling for the other treatment strategies)
2. 1 g of omega-3 fatty acids (EPA+DHA, ratio 1:2, from marine algae) compared to placebo (controlling for the other treatment strategies)
3. Home exercise program (muscle strength) of 30 minutes 3 times a week compared to a control exercise program (joint flexibility) 30 minutes 3 times a week

Follow-up: DO-HEALTH seniors will be followed for 3 years, in-person, and in 3-monthly intervals (4 clinical visits and 9 phone calls) at the 7 recruitment centers.

Study population: DO-HEALTH will enroll seniors age 70 years and older. To represent the largest part of the senior population, DO-HEALTH will recruit community-dwelling seniors. However, to represent also the pre-frail population at risk of institutionalization, at least 40% of seniors will be enrolled based on a fall with or without a fracture in the year before DO-HEALTH enrolment.

Study Design: This is a randomized, double-blind, placebo-controlled, 2×2×2 factorial design clinical trial.

Recruitment Centers: The trial will be performed at 7 recruitment centers located in 5 countries: Switzerland (University of Zurich, Basel University Hospital, Geneva University Hospital), France (University of Toulouse Hospital Centre), Germany (Charité Berlin), Portugal (University of Coimbra), and Austria (Innsbruck Medical University).

Randomization: Stratified block randomization. Labeling of study intervention will be performed by a central randomization centre in Switzerland.

Stratification variables: recruitment centre (7 centers), fall during previous 12 months (yes/no), gender, and age (70 - 84 and 85+). At least 40% of Seniors among those who fell or did not fall during the last year will be enforced at each of the 7 recruitment centers. Gender and age distribution will be monitored within each recruitment centre with the DO-HEALTH randomization software. If gross imbalance (less than 30% of fallers/non-fallers in a stratum) is detected within a centre, recruitment strategies for the centre will be adapted to boost recruitment of participants of underrepresented category.

website DO-HEALTH: http://do-health.eu/wordpress/

ELIGIBILITY:
Inclusion criteria:

* Age 70 years or older
* Mini Mental State Examination Score of at least 24
* Living in the community
* Sufficiently mobile to come to the study centre
* Able to walk 10 meters with or without a walking aid and able to get in and out of a chair without help
* Able to swallow study capsules
* Able and willing to participate, sign informed consent (including consent to analyze all samples until drop-out or withdrawal) and cooperate with study procedures

Exclusion criteria:

* Consumption of more than 1000 IU vitamin D/day in the 36 months prior to enrollment, or a bolus of 300'000 IU or more in the last 12 month prior to enrollment, and/ or unwillingness to limit vitamin D intake to the current standard of 800 IU/day of vitamin D during the course of the trial. Provision 1: an individual who consumed an average vitamin D dose between 1000 and 2000 IU vitamin D/day in the 3 months prior to enrollment, may be enrolled after a 3-month wash-out period where the maximum daily intake is limited to 800 IU vitamin D. Provision 2: an individual who consumed an average vitamin D dose higher than 2000 IU/day in the 3 months prior to enrollment, may be enrolled after a 6-month wash-out period where the maximum daily intake is limited to 800 IU vitamin D.
* Unwillingness to limit calcium supplement dose to 500 mg per day for the duration of the trial
* Taking omega-3 fat supplements in the 3 month prior to enrolment and unwilling to forgo their use for the duration of the trial
* Use of any active vitamin D metabolite (i.e. Rocaltrol, alphacalcidiol), PTH treatment (i.e. Teriparatide), or Calcitonin at baseline and unwillingness to forego these treatments during the course of the trial
* Current or recent (previous 4 months) participation in another clinical trial, or plans of such participation in the next 3 years (corresponding to DO-HEALTH length)
* Presence of the following diagnosed health conditions in the last 5 years: history of cancer (except non-melanoma skin cancer); myocardial infarction, stroke, transient ischemic attack, angina pectoris, or coronary artery intervention
* Severe renal impairment (creatinine clearance = 15 ml/min) or dialysis, hypercalcaemia (> 2.6 mmol/l)
* Hemiplegia or other severe gait impairment
* History of hypo- or primary hyperparathyroidism
* Severe liver disease
* History of granulomatous diseases (i.e. tuberculosis, sarcoidosis)
* Major visual or hearing impairment or other serious illness that would preclude participation
* Living with a partner who is enrolled in DO-HEALTH (i.e. only one person per household can be enrolled)
* Living in assisted living situations or a nursing home
* Temporary exclusion: acute fracture in the last 6 weeks
* Epilepsy and/or use of anti-epileptic drugs
* Individuals who fell more than 3 times in the last month
* Osteodystrophia deformans (M. Paget, Paget's disease)
* For study centers in Germany only: persons who are institutionalized / in prison by court order (§40, Abs. 1, Art. 4, "Gesetz über den Verkehr mit Arzneimitteln").

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2157 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Bone: Incident non-vertebral fractures over 36 months | over 36 months
  Confirmed by medical and/or x-ray reports
Muscle: Functional decline (lower extremity function) | Baseline, 12, 24 and 36 months
  Measured with the SPPB (short physical performance test battery)
Cardio-vascular: Systolic and diastolic blood pressure change | Baseline, 12, 24 and 36 months
  Standardized blood pressure assessment in sitting position
Brain: Cognitive decline | Baseline, 12, 24 and 36 months
  Montreal Cognitive Assessment (MoCA)
Immunity: Rate of any infections | Baseline, and every 3 months up to 36 months
  3-monthly incident infection protocol

SECONDARY OUTCOMES:
Bone: Incident hip fractures | 36 months
  Based on medical records and/or x-ray reports
Bone: Incident total fractures | 36 months
  Combined non-vertebral and vertebral fractures among subgroup of 1502 participants with DXA vertebral morphometry assessment
Bone: Incident vertebral fractures | 36 months
  Based on DXA vertebral morphometry among subset of 1502 participants
Bone: Bone mineral density decrease at the lumbar spine and hip | Baseline, 12, 24, and 36 months
  Assessed in a subset of 1502 participants with DXA measurements
Muscle: Rate of falls | Assessed every 3 months over 36 months
  Any low trauma fall, injurious fall
Muscle: reaction time and grip strength | Baseline, 12,24,36 months
  Reaction time will be assessed with the repeated sit-to-stand test; grip strength will be assessed with the Martin Vigorimeter
Muscle: Muscle mass decrease at upper and lower extremities | Baseline, 12,24,36 months
  Subset of 1502 participants with DXA measurements
Muscle: Dual tasking 10-meter gait speed | Baseline, 12,24 and 36 months
Muscle/Bone: musculoskeletal pain | Baseline, 12,24, and 36 months
  Assessed with the McGill questionnaire
Cardio-vascular: Incident Hypertension | 36 months
Brain: mental health decline | Baseline, 12,24, and 36 months
  Assessed with Geriatric Depression Scale
Brain: Incident Depression | 36 months
Brain/Muscle: Dual tasking gait variability | Baseline, 12, 24 and 36 months
  Subset of 250 participants
Immunity: Rate of upper respiratory infections / rate of flu-like illness | 36 months
  Assessed with infection protocol every 3 months
Immunity: Incident severe infections that lead to hospital admission | 36 months
Cartilage/Bone: Severity of knee pain in participants with symptomatic knee osteoarthritis | Baseline, 12, 24 and 36 months
  Assessed with the KOOS questionnaire. Knee OA assessment with modified ACR criteria.
Cartilage/Bone: Rate of knee buckling | Baseline, 12,24,36 months
  Questionnaire-based.
Cartilage/Bone: NSAID use / number of joints with pain | Baseline, 12, 24, 36 months
  Assessed by questionnaire and homunculus figure
Dental: Decline in oral health | Baseline, 12,24 and 36 months
  Assessed with questionnaire.
Dental: Tooth loss | 36 months
  Assessed by tooth count at every clinical visit
Gastro-Intestinal: rate of GI symptoms | Baseline, 12, 24 and 36 months
  Assessed with ROME III questionnaire.
Glucose-Metabolic: Change in fasting glucose, insulin levels (QUICKI, HOMA index) | Baseline, 12,24,36 months
  Laboratory measures at the Central DO-HEALTH Laboratory (Institute of Clinical Chemistry at the University Hospital Zurich)
Glucose-Metabolic: Body composition | Baseline, 12, 24, 36 months
  Subset of 1502 participants with DXA measurements
Kidney: Decline in kidney function | Baseline, 12, 24, and 36 months
  Blood creatinine levels and estimated glomerular filtration rate
Global Health: Quality of life | Every 6 months
  Assessed with questionnaire (EuroQuol).
Global Health: Incident disability regarding activities of daily living | Baseline, 12, 24 and 36 months
  Assessed with HAQ-PROMIS questionnaire
Global Health: Incident nursing home admission | 36 months
Global Health: Mortality | 36 months

OTHER OUTCOMES:
Biomarker endpoints | Baseline, 12, 24, and 36 months
Bone: Incident repeat fractures | 36 months
  Any repeat non-vertebral fractures in all participants, vertebral fractures and total fractures among subset of 1502 seniors with yearly DXA measurements
BONE: Functional recovery after long bone fracture | 36 months
Muscle: Incident sarcopenia / incident frailty / decline in physical function | 36 months
  Incident sarcopenia (among subset of 1502 seniors with yearly DXA measurements), incident frailty (questionnaire), decline in physical activity (questionnaire)
Cardio-vascular: Major cardio-vascular events | 36 months
  Major cardiovascular events as a composite endpoint (any event: myocardial infarction, stroke, revascularization procedures of CABG and PCI, incident congestive heart disease, cardiovascular mortality); individual endpoints: myocardial infarction, stroke, incident congestive heart disease, and cardiovascular mortality (assessed every 3 months over 36 months)
Brain: incident dementia | 36 months
Immunity: Incident cancer / rate of implant infections / rate of gastro-intestinal infections | 36 months
  Incident cancer (any cancer, gastro-intestinal, breast cancer in women, prostate cancer in men); rate of implant infections after total hip or knee replacement (due to fracture or osteoarthritis); rate of gastro-intestinal infections
Cartilage/bone: Incident osteoarthritis | Baseline, 12, 24, and 36 months
  Incident symptomatic knee osteoarthritis; incident symptomatic hip osteoarthritis, incident symptomatic hand osteoarthritis; composite endpoint: incident symptomatic knee, hip or hand osteoarthritis; severity of hip pain in those with prevalent symptomatic hip osteoarthritis, severity of hand pain in those with prevalent symptomatic hand osteoarthritis
Adherence laboratory | Baseline, 12, 24, and 36 months
  Serum 25(OH)D concentrations (measured both by an automated assay and HPLCMS/MS) and plasma PUFA concentrations (EPA, AA, DPA, DHA; measured by a sensitive and selective assay based on gas chromatography coupled to mass spectrometry detection (GC-MS)) in all participants

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff Ferrari, Prof MD, Principal Investigator — "Centre on Aging and Mobility" University of Zurich, University Hospital Zurich and City Hospital Waid.
Locations (7):
- University of Innsbruck, Innsbruck, Austria
- University of Toulouse - Centre de Recherche - Gérontopôle Hôpital La Grave, Toulouse, France
- Charité Berlin, Berlin, Germany
- University of Coimbra - Clínica Universitária de Reumatologia, Coimbra, Portugal
- Switzerland (3):
  - Centre on Aging and Mobility, University of Zurich and City Hospital Waid, Zurich, Canton of Zurich
  - Basel University, Basel
  - Hôpitaux Universitaires de Genève, Geneva

REFERENCES:
- [Derived] Wieczorek M, Funk J, Mattle M, Gangler S, Egli A, Kressig RW, Manz MG, Bischoff-Ferrari HA; DO-HEALTH Research group. Association between hemoglobin levels and mild cognitive impairment in generally healthy European community-dwelling older adults: a 3-year prospective analysis of the DO-HEALTH trial. Am J Clin Nutr. 2025 Nov 13:101114. doi: 10.1016/j.ajcnut.2025.11.005. Online ahead of print. PMID 41241003
- [Derived] Kistler-Fischbacher M, Gohar G, de Godoi Rezende Costa Molino C, Geiling K, Meyer-Heim T, Kressig RW, Orav EJ, Vellas B, Guyonnet S, da Sliva JAP, Rizzoli R, Armbrecht G, Steinhagen-Thiessen E, Egli A, Bischoff-Ferrari HA. Cognitive function in generally healthy adults age 70 years and older in the 5-country DO-HEALTH study: MMSE and MoCA scores by sex, education and country. Aging Clin Exp Res. 2025 Mar 17;37(1):88. doi: 10.1007/s40520-025-02946-4. PMID 40095212
- [Derived] de Godoi Rezende Costa Molino C, Forster CK, Wieczorek M, Orav EJ, Kressig RW, Vellas B, Egli A, Freystaetter G, Bischoff-Ferrari HA; DO-HEALTH Research Group. Association of fall risk-increasing drugs with falls in generally healthy older adults: a 3-year prospective observational study of the DO-HEALTH trial. BMC Geriatr. 2024 Nov 29;24(1):980. doi: 10.1186/s12877-024-05557-2. PMID 39614147
- [Derived] Gaengler S, Sadlon A, De Godoi Rezende Costa Molino C, Willett WC, Manson JE, Vellas B, Steinhagen-Thiessen E, Von Eckardstein A, Ruschitzka F, Rizzoli R, da Silva JAP, Kressig RW, Kanis J, Orav EJ, Egli A, Bischoff-Ferrari HA. Effects of vitamin D, omega-3 and a simple strength exercise programme in cardiovascular disease prevention: The DO-HEALTH randomized controlled trial. J Nutr Health Aging. 2024 Feb;28(2):100037. doi: 10.1016/j.jnha.2024.100037. Epub 2024 Jan 9. PMID 38199870
- [Derived] Gagesch M, Wieczorek M, Abderhalden LA, Lang W, Freystaetter G, Armbrecht G, Kressig RW, Vellas B, Rizzoli R, Blauth M, Orav EJ, Egli A, Bischoff-Ferrari HA. Grip strength cut-points from the Swiss DO-HEALTH population. Eur Rev Aging Phys Act. 2023 Aug 5;20(1):13. doi: 10.1186/s11556-023-00323-6. PMID 37543639
- [Derived] Bischoff-Ferrari HA, Willett WC, Manson JE, Dawson-Hughes B, Manz MG, Theiler R, Braendle K, Vellas B, Rizzoli R, Kressig RW, Staehelin HB, Da Silva JAP, Armbrecht G, Egli A, Kanis JA, Orav EJ, Gaengler S. Combined Vitamin D, Omega-3 Fatty Acids, and a Simple Home Exercise Program May Reduce Cancer Risk Among Active Adults Aged 70 and Older: A Randomized Clinical Trial. Front Aging. 2022 Apr 25;3:852643. doi: 10.3389/fragi.2022.852643. eCollection 2022. PMID 35821820
- [Derived] de Godoi Rezende Costa Molino C, Chocano-Bedoya PO, Sadlon A, Theiler R, Orav JE, Vellas B, Rizzoli R, Kressig RW, Kanis JA, Guyonnet S, Lang W, Egli A, Bischoff-Ferrari HA; DO-HEALTH Research Group. Prevalence of polypharmacy in community-dwelling older adults from seven centres in five European countries: a cross-sectional study of DO-HEALTH. BMJ Open. 2022 Apr 29;12(4):e051881. doi: 10.1136/bmjopen-2021-051881. PMID 35487733
- [Derived] Schietzel S, Chocano-Bedoya PO, Sadlon A, Gagesch M, Willett WC, Orav EJ, Kressig RW, Vellas B, Rizzoli R, da Silva JAP, Blauth M, Kanis JA, Egli A, Bischoff-Ferrari HA. Prevalence of healthy aging among community dwelling adults age 70 and older from five European countries. BMC Geriatr. 2022 Mar 2;22(1):174. doi: 10.1186/s12877-022-02755-8. PMID 35236290
- [Derived] Bischoff-Ferrari HA, Vellas B, Rizzoli R, Kressig RW, da Silva JAP, Blauth M, Felson DT, McCloskey EV, Watzl B, Hofbauer LC, Felsenberg D, Willett WC, Dawson-Hughes B, Manson JE, Siebert U, Theiler R, Staehelin HB, de Godoi Rezende Costa Molino C, Chocano-Bedoya PO, Abderhalden LA, Egli A, Kanis JA, Orav EJ; DO-HEALTH Research Group. Effect of Vitamin D Supplementation, Omega-3 Fatty Acid Supplementation, or a Strength-Training Exercise Program on Clinical Outcomes in Older Adults: The DO-HEALTH Randomized Clinical Trial. JAMA. 2020 Nov 10;324(18):1855-1868. doi: 10.1001/jama.2020.16909. PMID 33170239
- See also: European Commission project link for DO-HEALTH — http://ec.europa.eu/research/health/medical-research/human-development-and-ageing/projects/do-health_en.html
- See also: Website DO-HEALTH Consortium — http://do-health.eu